CLINICAL TRIAL: NCT07003490
Title: Radical Resection With Contralateral Lymph Node Dissection in Clinical Stage N3 Non-Small Cell Lung Cancer
Brief Title: Radical Resection With Contralateral Lymph Node Dissection for Clinical N3 NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Wu Liang, Associate Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025HS068
Record Dates: First submitted 2025-04-18; First posted 2025-06-04 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: NSCLC, Non Small Cell Lung Cancer
Keywords: NSCLC; Lung cancer; Lymph node dissection; Radical resection; Surgery; N3 stage; Stage IIIB; Contralateral lymph node metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: single center, single arm, interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical treatment group (Experimental): Patients in this arm are diagnosed with clinical N3 stage lung cancer which specifically involves contralateral lymph node metastasis by PET scan. And these patients will be treated with radical resection with bilateral lymph node dissection.
  Interventions: Procedure: Radical Resection with Bilateral Lymph Node Dissection

INTERVENTIONS:
Procedure: Radical Resection with Bilateral Lymph Node Dissection — The patient will be positioned in a contralateral decubitus position based on the location of the primary tumor, with the axillary region on the side of the primary tumor exposed. For example, if the patient is diagnosed with left-sided primary lung cancer with right-sided lymph node metastasis, investigators perform left axillary incision to resect the tumor. And then investigators change the patient's position to perform right axillary incision to resect the lymph nodes. Thoracoscopy surgery will be used to access and resect the primary lesion and lymph node metastasis.

SUMMARY:
*Study Overview This study is investigating a surgical approach for patients with a serious type of lung cancer known as non-small cell lung cancer (NSCLC), particularly those in an advanced stage where cancer has spread to both sides of the chest (referred to as N3 stage). In these patients, the cancer has spread to contralateral lymph nodes, which are lymph nodes located on the opposite side of the chest. This spread makes the cancer harder to treat and lowers the chance of survival.

The study is focusing on whether removing the primary lung tumor along with lymph nodes from both sides of the chest-a surgery called bilateral lymph node dissection-can improve the chances of survival and reduce the risk of cancer returning.

*Why This Study Is Important Stage N3 NSCLC (where cancer has spread to both sides of the chest) is hard to treat and has a poor prognosis. Current treatments include surgery, chemotherapy, and radiation, but the long-term survival rates are still low.

This study will evaluate whether surgery alone (with the tumor and lymph nodes removed) can improve survival in these patients compared to other treatment options.

The goal is to find the best way to treat patients with N3 stage NSCLC by studying the risks and benefits of this combined surgical approach.

* What the Study Is Testing

  1. Effectiveness of surgery for N3 stage patients: Does removing both the primary tumor and lymph nodes from both sides of the chest improve survival rates?
  2. Safety of the surgery: What are the risks or complications from such an extensive operation? For example, the study will check for things like infections, lung function problems, and other side effects.
  3. Impact of other treatments: The study will also look at whether treatments like chemotherapy or radiation before surgery (called neoadjuvant therapy) change the results of surgery.
  4. Impact of lymph node involvement: The study will examine how many lymph nodes are affected by cancer and how this affects treatment outcomes.
* Who Can Participate? The study is looking for people diagnosed with N3 stage NSCLC, meaning their cancer has spread to lymph nodes on both sides of the chest. Patients must be considered eligible for surgery based on their overall health and the specific characteristics of their cancer.
* What Will the Patients Experience? Patients who take part in this study will undergo surgery to remove their lung tumor and lymph nodes from both sides of the chest.

They will receive follow-up care to monitor for any complications, such as infections, and to see if the cancer comes back.

Patients will be monitored for several years to track their survival, recurrence of cancer, and any long-term effects of the surgery.

*What Could This Mean for Patients? If the study shows that this combined surgery approach is effective, it could become a standard treatment for patients with N3 stage NSCLC, improving their chances of survival and possibly reducing the need for more aggressive treatments like chemotherapy or radiation in the future.

However, it's important to note that surgery of this type comes with risks, and not all patients will be suitable candidates for this approach. The study aims to better understand these risks and benefits to help doctors make the best treatment decisions for each individual patient.

*Key Takeaways for Healthcare Providers The study is investigating radical surgery for N3 stage NSCLC, with an emphasis on bilateral lymph node dissection to improve survival.

The study will assess surgical outcomes, complications, and long-term survival rates in patients with metastasis to lymph nodes on both sides of the chest.

Findings may lead to a new approach in treating patients with N3 stage lung cancer, offering potential improvements in patient outcomes.

DETAILED DESCRIPTION:
1. Background Lung cancer is one of the most common malignant tumors worldwide and a leading cause of cancer-related mortality. According to cancer statistics, approximately 1.8 million people die from lung cancer annually worldwide. In China, the incidence and mortality rates of lung cancer are on the rise, particularly for non-small cell lung cancer (NSCLC), which accounts for approximately 85% of all lung cancer cases. Many lung cancer patients already present with contralateral mediastinal or hilar lymph node metastasis at the time of diagnosis, which corresponds to N3 stage in lymph node staging. N3 stage lung cancer is classified as locally advanced or metastatic disease. Due to its aggressive progression and extensive invasiveness, clinical diagnosis and treatment of N3 stage lung cancer pose significant challenges. Therefore, effectively assessing lymph node metastasis in lung cancer patients and developing personalized treatment strategies for those with contralateral thoracic lymph node metastasis has become a central topic in clinical research.

   The staging system for lung cancer is based on tumor size, lymph node involvement, and the presence of distant metastasis. According to the eighth edition of the TNM staging system released by the International Association for the Study of Lung Cancer (IASLC), lymph node metastasis (N stage) is a core factor in determining prognosis and treatment decisions. N stage not only assesses whether the tumor has spread to adjacent lymph nodes, but also includes the specific location and number of affected nodes. N0 indicates no lymph node metastasis, N1 indicates metastasis to proximal hilar lymph nodes, N2 indicates metastasis to mediastinal lymph nodes, and N3 indicates distant lymph node metastasis, which typically involves contralateral thoracic lymph nodes and cervical lymph nodes. N3 stage lung cancer is usually considered as locally advanced or metastatic disease, with a poor prognosis. The 1-year, 3-year, and 5-year overall survival rates are 35.8%, 6.8%, and 1.7%, respectively, while the corresponding cancer-specific survival rates are 36.6%, 6.9%, and 1.8%. Contralateral thoracic lymph node metastasis is a specific type of N3 stage lymph node metastasis, indicating that cancer cells have spread from the primary tumor to the contralateral thoracic lymph nodes through the lymphatic system. The presence of contralateral thoracic lymph node metastasis usually signifies that cancer has crossed the midline of the thoracic cavity, increasing the cancer's invasiveness and the complexity of surgical treatment. For clinically staged N3 NSCLC patients, treatment strategies often require a combination of surgery, radiotherapy, chemotherapy, and chemoradiotherapy to improve survival and control symptoms. However, due to the presence of contralateral thoracic lymph node metastasis, surgical resection alone is often insufficient for achieving optimal cure, and lymph node dissection becomes an indispensable part of the treatment plan.

   Currently, treatment strategies for N3 stage lung cancer with contralateral thoracic lymph node metastasis emphasize multimodal approaches. Traditional treatment options include surgery, chemotherapy, radiotherapy, and chemoradiotherapy combinations, aiming to improve survival rates and control symptoms. In recent years, targeted therapies and immunotherapies have also been increasingly applied in the treatment of N3 stage lung cancer, offering new hope for patients who were previously considered unsuitable for surgery or with limited treatment options. Immunotherapy, particularly immune checkpoint inhibitors, has been used as a first-line treatment for metastatic disease and as consolidation therapy after chemoradiotherapy for unresectable locally advanced disease. Targeted therapies have improved prognosis for patients with specific genetic mutations (e.g., EGFR mutations and ALK rearrangements). These therapies are personalized based on the tumor's molecular characteristics, representing a more individualized approach to treatment. However, the development of resistance to these therapies by tumor cells remains an unresolved issue. The combination of immunotherapy in N3 stage NSCLC has improved surgical success rates and reduced postoperative recurrence. However, the side effects of immunotherapy significantly limit its widespread application in lung cancer. Surgery remains the primary treatment for early-stage lung cancer, but due to the extensive lymph node metastasis in N3 stage patients, the difficulty of lymph node dissection increases, and guidelines do not recommend primary surgery for N3 stage lung cancer patients.

   Management of N3 stage NSCLC remains controversial due to the heterogeneity of the disease and the limited efficacy of current treatment methods. For patients with contralateral thoracic lymph node metastasis, the suitability of surgery remains a topic of debate. On one hand, surgical resection can significantly improve local control rates, particularly in patients who are amenable to resection. A retrospective analysis of N3 stage lung cancer patients found that lobectomy combined with lymph node dissection could improve overall survival and local control rates compared to non-surgical treatments. Additionally, Bott et al. reported that N3 stage lung cancer patients who underwent surgical resection had a higher median overall survival (OS) compared to those who did not undergo surgery. On the other hand, the widespread and multifocal nature of lymph node metastasis in N3 stage patients requires an expanded surgical resection to achieve complete removal of the tumor and affected lymph nodes, significantly increasing the complexity and risk of surgery.

   Although surgical treatment for N3 stage lung cancer with contralateral thoracic lymph node metastasis has been relatively rare, bilateral lymph node dissection has been consistently regarded as an important component of surgery for N3 stage patients, especially those with contralateral thoracic lymph node metastasis. Bilateral lymph node dissection not only helps to remove the tumor and its metastases more thoroughly but also improves the lymph node clearance rate, thereby reducing the risk of postoperative recurrence. Riquet et al. retrospectively analyzed 11 pN3 patients, all of whom underwent complete resection of the primary tumor and ipsilateral mediastinal lymph node dissection. Seven of them also underwent additional N3 lymph node dissection, and four of these patients were alive at five years of follow-up with good survival outcomes. Another retrospective study analyzed 11 N3 stage lung cancer patients who underwent bilateral lymph node dissection. Among those with left-sided lung cancer, six patients had a 100% five-year survival rate, while five right-sided lung cancer patients had a 30% three-year survival rate. Hata et al. reported a high five-year survival rate (62.5%) with conventional thoracotomy combined with bilateral lymph node dissection in eight N3 stage lung cancer patients. Furthermore, Watanabe et al. employed median sternotomy to perform extensive bilateral hilar, mediastinal, and supraclavicular lymph node dissection in 19 N3 stage lung cancer patients, with six patients still alive at the end of the study, and the longest survival time was 23 months, although the longest follow-up period in this study was less than five years.

   Currently, research on the application of primary surgical interventions in clinically staged N3 NSCLC patients remains limited, with most studies being retrospective analyses with small sample sizes. The existing studies show significant heterogeneity in surgical techniques and lymph node dissection strategies, making it difficult to discern the specific differences in efficacy between different surgical approaches and lymph node dissection methods for N3 stage lung cancer. Additionally, many related studies are relatively old, with lymph node dissection techniques mainly involving median sternotomy for bilateral thoracic lymph node dissection. This technique, being more invasive, may adversely affect postoperative recovery and survival outcomes for patients.

   In recent years, with the rapid development of thoracoscopic technology, the invasiveness of lung cancer surgery has been significantly reduced, leading to improved postoperative recovery, reduced complications, and better quality of life for patients. Thoracoscopic surgery not only achieves higher R0 resection rates but also effectively improves local tumor control, especially in handling N3 stage lymph node metastasis. Therefore, with ongoing advancements in surgical techniques and postoperative care, the treatment approach of primary tumor resection combined with bilateral lymph node dissection may offer less surgical trauma, higher complete resection rates, and significant improvements in local control and survival for patients with locally advanced lung cancer.

   N3 stage lung cancer with contralateral thoracic lymph node metastasis presents a complex and challenging clinical problem. Although bilateral lymph node dissection has shown positive results in some patients, its high-risk profile and complications in previous studies raise questions about whether primary surgical intervention can be expanded to more N3 stage patients. Minimally invasive lung tumor resection surgery offers a promising approach to controlling locally advanced lung cancer and improving patient survival.
2. Purpose

   Primary Purpose:

   - Evaluate the efficacy of primary tumor resection combined with bilateral lymph node dissection in non-small cell lung cancer (NSCLC) patients with contralateral thoracic lymph node metastasis detected by PET: The primary objective is to assess the clinical efficacy of primary tumor resection combined with bilateral lymph node dissection in terms of postoperative survival rates (such as overall survival and disease-free survival).

   Secondary Purpose:

   - Investigate the impact of primary tumor resection combined with bilateral lymph node dissection on postoperative complications: This objective aims to evaluate the potential complications arising from the surgical procedure, including postoperative infection, lymphatic leakage, respiratory dysfunction, and atrial fibrillation, as well as analyze the safety of this combined surgical approach.

   - Assess the extent of surgical trauma caused by primary tumor resection combined with bilateral lymph node dissection: The study will examine key indicators of surgical trauma, such as intraoperative blood loss, postoperative pain scores, and length of hospital stay, to provide evidence for the safety and feasibility of this combined treatment approach and offer guidance for postoperative management and patient recovery optimization.
   * Analyze the impact of neoadjuvant therapy on the efficacy of primary tumor resection combined with bilateral lymph node dissection: This objective aims to explore the effects of neoadjuvant therapy (or the lack thereof) and different neoadjuvant treatment regimens on patient survival, recurrence rates, and postoperative complications, in order to identify key factors that may influence treatment outcomes.
   * Evaluate the impact of lymph node metastasis during lymph node dissection and its prognostic predictive value: This objective will analyze the effect of the number and location of lymph node metastases on patient prognosis, as well as assess the benefit-risk ratio of applying this combined therapy in patients who are pathologically classified as non-N3 (i.e., those without contralateral thoracic lymph node metastasis).
3. Study Design

   - Study Type This study is a single-center, prospective, single-arm trial. The primary objective of the study is to evaluate the efficacy of primary tumor resection combined with bilateral lymph node dissection in non-small cell lung cancer (NSCLC) patients with contralateral thoracic lymph node metastasis detected by PET. The study will also assess the surgical trauma and the impact of neoadjuvant therapy on treatment outcomes. Furthermore, the study will explore the impact of the number and location of lymph node metastasis on prognosis, as well as the benefit-risk ratio of this treatment approach in patients who are pathologically classified as non-N3 (i.e., without contralateral thoracic lymph node metastasis) based on postoperative pathological examination.

   Subjects enrolled in the study will be diagnosed with primary tumors accompanied by contralateral lymph node metastasis based on PET scan results. After preoperative evaluation and exclusion of any surgical contraindications, these patients will undergo scheduled surgery. Postoperatively, the patients will be followed up to observe their survival outcomes (such as overall survival and disease-free survival) to assess the clinical efficacy of the treatment. The study will evaluate the safety and effectiveness of the treatment through various indicators, including surgical duration, incision size, surgical difficulty, intraoperative blood loss, postoperative drainage, complication rates, and length of hospitalization.

   For patients with postoperative pathological examination indicating non-contralateral thoracic lymph node metastasis (non-pathological N3 stage), a subgroup analysis will be conducted to compare their prognosis with patients who have the same N stage and baseline characteristics but who did not receive surgical treatment. This will allow for the evaluation of the benefit-risk ratio of the treatment for this subgroup of patients. Statistical analysis will be independently conducted by designated statistical experts.
   * Sample Size Estimation The study will include untreated NSCLC patients who have been diagnosed through clinical imaging (PET or contrast-enhanced CT) with primary tumors and contralateral lymph node metastasis. A total of 30 patients meeting the inclusion criteria are expected to be enrolled during the study period. The sample size was determined considering the study design, effect size, statistical power, and operational feasibility in clinical practice to ensure the scientific rigor and reliability of the results.
   * Study Site The study will be conducted at the Department of Thoracic Surgery, Shanghai First People's Hospital.
   * Study Implementation Patients will be enrolled in the study after their preoperative PET scan confirms primary tumors with contralateral thoracic lymph node metastasis, and after communication with the patients and their families regarding consent for participation. Enrolled patients will undergo preoperative evaluation and, following the exclusion of surgical contraindications, will undergo scheduled surgery.

   The study will evaluate the safety and effectiveness of the combined treatment approach using various indicators such as surgical time, incision size, surgical difficulty, intraoperative blood loss, postoperative drainage, complication rates, and recovery time. A subgroup analysis will be performed comparing non-pathological N3 patients (those without contralateral thoracic lymph node metastasis) with patients who have the same N stage and baseline characteristics but who received non-surgical intervention. This will assess the benefit-risk ratio of the treatment for this subgroup of patients.
4. Follow-up Plan

   To ensure postoperative recovery, assess the surgical outcomes, and monitor for potential recurrence, all enrolled patients will undergo regular follow-up assessments as part of this study. The follow-up plan will include the following components:
   * Follow-up Frequency and Schedule 1 Month Postoperatively: The first follow-up will primarily assess postoperative recovery, including physical condition, changes in symptoms, and the occurrence of any postoperative complications.

     3 Months Postoperatively: The follow-up will evaluate tumor recurrence or metastasis, including chest imaging (such as chest CT or PET-CT) and necessary blood tests (such as tumor markers).

     6 Months Postoperatively: The follow-up will include imaging and tumor marker testing, focusing on any new tumor lesions or signs of recurrence.

   Annually Postoperatively: Long-term follow-up will continue to monitor survival status, quality of life, tumor recurrence, and potential late-term complications.
   * Follow-up Components

     1. Clinical Assessment: This will include routine physical examinations, symptom evaluations (e.g., cough, dyspnea, chest pain), and quality of life questionnaires.
     2. Imaging: All patients will undergo chest CT or PET-CT scans at the 1-month, 3-month, and 6-month follow-up visits, as well as annually thereafter, to assess tumor recurrence, metastasis, and other relevant pathologies.
     3. Laboratory Tests: Blood tests will be conducted at the 1-month, 3-month, and 6-month follow-ups, focusing on tumor markers (such as CEA), as well as routine blood counts, liver and kidney function tests, and inflammatory markers.
     4. Lymph Node Monitoring: Throughout the follow-up process, lymph nodes in the thoracic and other relevant areas will be dynamically monitored to detect any early signs of metastatic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary non-small cell lung cancer (NSCLC): The diagnosis must be confirmed through pathological examination, and the patient must meet one of the following histological types: adenocarcinoma, squamous cell carcinoma, or large cell carcinoma.
* PET-CT indicating contralateral mediastinal lymph node metastasis, N3 stage: Patients must have lung cancer classified as stage N3 based on positron emission tomography (PET) scans, with evidence of contralateral mediastinal lymph node involvement.
* Age range: Patients must be aged between 18 and 75 years.
* Good cardiopulmonary function:Preoperative evaluation must show no significant cardiovascular conditions (e.g., heart failure, severe coronary artery disease) or severe respiratory diseases (e.g., chronic obstructive pulmonary disease), and the patient must have good heart function (LVEF ≥ 45%), with the ability to tolerate surgery.Preoperative pulmonary function assessment must meet the surgical criteria, with forced expiratory volume in 1 second (FEV1) ≥ 50% of predicted value.
* Resectable tumor: Based on imaging studies (such as CT or MRI) and assessment by thoracic surgeons, the patient must be deemed suitable for surgical resection and planned for primary tumor resection combined with bilateral lymph node dissection.
* No distant metastasis: Full-body imaging (such as CT or PET-CT) must show no evidence of distant metastasis, indicating that the patient is suitable for localized treatment.
* ECOG performance status of 0-1: Patients must have an ECOG performance status score of 0-1 (as per Attachment 1), indicating that they are clinically in good physical condition and able to perform daily activities independently.
* Informed consent: The patient and their family members must voluntarily sign an informed consent form after being fully informed of the purpose, content, risks, and potential benefits of the study, consenting to participate in the research.

Exclusion Criteria:

* Patients with unresectable tumors: This includes patients with tumors extensively invading vital organs (e.g., major blood vessels, spine, heart) or those for whom complete surgical resection is not feasible.
* Patients with severe comorbidities: These include individuals with severe cardiovascular diseases (e.g., heart failure, history of myocardial infarction, arrhythmia), severe respiratory diseases (e.g., chronic obstructive pulmonary disease, severe asthma), or other uncontrolled systemic diseases that may affect the patient's ability to tolerate surgery safely.
* Patients with distant metastasis: This includes patients with imaging findings suggestive of metastasis to distant organs, such as the liver, bones, or brain.
* Patients with allergies to anesthetic agents or contraindications to anesthesia: This includes patients with a history of severe allergies or those with significant pulmonary or cardiovascular comorbidities that increase the anesthesia risk.
* Pregnant or lactating women: Due to potential risks associated with radiological examinations (e.g., PET scans) and surgery for the fetus or infant.
* Patients with psychiatric disorders or those unable to comprehend the informed consent form: This includes patients who are unable to provide independent informed consent or fully understand the study protocol and associated risks.
* Patients unable to comply with follow-up requirements: This includes patients who are unable to attend scheduled postoperative follow-up visits, such as those living far from the hospital or with other logistical barriers.
* Patients with concurrent malignant hematologic diseases or other primary cancers: This includes patients who have other primary malignancies, especially those with high recurrence risks, in addition to lung cancer.
* Patients with known immune deficiencies or immune system disorders: This includes patients with severe immunodeficiency diseases, HIV, a history of organ transplantation, or other conditions that may compromise postoperative recovery and affect the efficacy of antitumor treatments.
* Elderly patients unable to tolerate surgery or anesthesia: This includes elderly individuals with multiple chronic conditions or functional decline, making them unable to tolerate surgical risks.
* Patients with severe hepatic or renal dysfunction: This includes patients with liver cirrhosis, renal failure, or other severe organ dysfunction that may prevent them from tolerating surgery and postoperative treatments.
* Patients with active infections: This includes patients with active infectious diseases, such as pneumonia being treated with antibiotics, especially those with contagious conditions such as tuberculosis or bacterial pneumonia.
* Patients with severe diabetes: This includes patients with unstable blood sugar control and diabetes-related complications (e.g., diabetic retinopathy, diabetic foot) that may complicate postoperative recovery.
* Patients currently participating in other clinical trials: This includes patients enrolled in other clinical studies whose treatments may interfere with the interventions in this study.
* Patients with severe malnutrition: This includes patients with significant weight loss or malnutrition that may impair postoperative recovery and increase anesthesia risk.
* Patients with severe hematological disorders: This includes patients with conditions such as anemia or thrombocytopenia, which could complicate hemostasis during surgery and postoperative recovery.
* Patients with severe chronic respiratory failure: This includes patients who are long-term ventilator-dependent or require tracheostomy, as they may have a higher surgical risk and compromised postoperative recovery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Efficacy of Primary Tumor Resection Combined with Bilateral Lymph Node Dissection in Non-Small Cell Lung Cancer Patients with Contralateral Thoracic Lymph Node Metastasis | 12 months for disease-free survival
  The clinical efficacy of the surgery in contralateral lymph node metastasis patients will be assessed by analyzing postoperative disease-free survival (DFS).

SECONDARY OUTCOMES:
Evaluation of intra-operative blood loss | Perioperative
  Intra-operative blood loss volume (ml) recored during operation will be one of the parameters to evaluate safety of the surgery
Evaluation of post-operative pain | Perioperative
  Post-operative pain scores recorded by Visual Analogue Scale (higher sores indicate more severe pain) will be one of the parameters to evaluate tolerability of the surgery
Evaluation of incidence of post-operative complications | Perioperative
  Incidence of post-operative complications such as pleural effusion, recurrent laryngeal nerve injury and arrhythmia will be one of the parameters to evaluate safety and tolerability of the surgery.
Evaluation of chest tube retention time | Perioperative
  Chest tube retention time (days) will be one of the parameters to evaluate surgical trauma
Evaluation of chest tube drainage output | Perioperative
  Chest tube drainage output (ml) will be one of the parameters to evaluate surgical trauma
The impact of neoadjuvant therapy on the safety of surgery | Perioperative/Periprocedural
  Analyze the impact of preoperative use or non-use of neoadjuvant therapy, as well as different neoadjuvant therapy regimens, postoperative complications
The impact of neoadjuvant therapy on the efficacy of surgery | Disease-free survival rate at 12 months post operative for the analyzation of patient survival and recurrence rates.
  Analyze the impact of preoperative use or non-use of neoadjuvant therapy, as well as different neoadjuvant therapy regimens, on patient recurrence rates.
Evaluation of the impact of lymph node metastasis on surgical outcomes | 12 months for disease-free survival
  Investigate the impact of the number and location of lymph node metastasis on surgical outcomes and patient prognosis.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai General Hospital Thoracic Surgery Department, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Watanabe Y, Shimizu J, Oda M, Hayashi Y, Tatsuzawa Y, Watanabe S, Urayama H, Iwa T. Results of surgical treatment in patients with stage IIIB non-small-cell lung cancer. Thorac Cardiovasc Surg. 1991 Feb;39(1):50-4. doi: 10.1055/s-2007-1013930. PMID 1849325
- [Background] Beck SL. Prenatal and postnatal assessment of Maneb-exposed CD-1 mice. Reprod Toxicol. 1990;4(4):283-90. doi: 10.1016/0890-6238(90)90040-3. PMID 2136049
- [Background] Bott MJ, Patel AP, Crabtree TD, Morgensztern D, Robinson CG, Colditz GA, Waqar S, Kreisel D, Krupnicka AS, Patterson GA, Broderick S, Meyers BF, Puri V. Role for Surgical Resection in the Multidisciplinary Treatment of Stage IIIB Non-Small Cell Lung Cancer. Ann Thorac Surg. 2015 Jun;99(6):1921-8. doi: 10.1016/j.athoracsur.2015.02.033. Epub 2015 Apr 23. PMID 25912748
- [Background] Tian Z, Zhang J, Liu D, Liang C. Lobectomy with Lymph Node Dissection Benefits N3 Stage Non-Small Cell Lung Cancer Patients: A Population-Based Study. Oncology. 2025;103(6):445-455. doi: 10.1159/000541634. Epub 2024 Sep 30. PMID 39348811
- [Background] Riquet M, Mordant P, Fabre-Guillevin E, Arame A, Foucault C, Dujon A, Le Pimpec Barthes F. Long-term survival with surgery as part of a multimodality approach for N3 lung cancer. Eur J Cardiothorac Surg. 2013 Dec;44(6):1117-22. doi: 10.1093/ejcts/ezt171. Epub 2013 Mar 29. PMID 23543202